CLINICAL TRIAL: NCT00917644
Title: An Open Label, Randomized, Single Dose, Two-Way Crossover Bioequivalence Study Comparing A New 80 Mg Atorvastatin Tablet To A 80 Mg Atorvastatin Commercial Tablet In Healthy Subjects
Brief Title: Bioequivalence Study Comparing A New 80 Mg Atorvastatin Tablet To A 80 Mg Atorvastatin Commercial Tablet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A2581167
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Results first posted 2009-10-15 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: Bioqeuivalence, Pharmacokinetics, Atorvastatin
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Other): 80 mg atorvastatin tablets
  Interventions: Drug: Atorvastatin
- Test (Experimental): New 80 mg atorvastatin tablets
  Interventions: Genetic: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — A single 80 mg dose of marketed 80 mg atorvastatin tablets
  Arms: Reference
Genetic: Atorvastatin — A single dose of new formulation of 80 mg atorvastatin tablets
  Arms: Test

SUMMARY:
To determine whether new 80 mg atorvastatin tablets are bioequivalent to 80 mg commercial atorvastatin tablets (Lipitor®).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 18 to 30 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.
* Treatment with an investigational drug within 30 days or 5 half lives preceding the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581167&StudyName=Bioequivalence%20Study%20Comparing%20A%20New%2080%20Mg%20Atorvastatin%20Tablet%20To%20A%2080%20Mg%20Atorvastatin%20Commercial%20Tablet

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Drug First: New (test) 80 milligram (mg) atorvastatin tablets as a single dose in the first intervention period and marketed (reference) 80 mg atorvastatin commercial tablet (Lipitor®) as a single dose in the second intervention period (after washout period).
- Reference Drug First: Marketed (reference) 80 mg atorvastatin commercial tablet (Lipitor®) as a single dose in the first intervention period and new (test) 80 mg atorvastatin tablets as a single dose in the second intervention period (after washout period).
Period: Period 1: First Intervention
Arm/Group | Test Drug First | Reference Drug First
Started | 39 | 37
Completed | 39 | 37
Not Completed | 0 | 0
Period: Period: Washout Period of > = 2 Weeks
Arm/Group | Test Drug First | Reference Drug First
Started | 39 | 37
Completed | 37 | 37
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2: Second Intervention
Arm/Group | Test Drug First | Reference Drug First
Started | 37 (Washout: Test drug 1st, completed = 37; 2nd period: Test drug 2nd, completed = 37.) | 37 (Washout: Reference drug (Ref) 1st, completed = 37; 2nd period: Ref drug 2nd, completed = 36.)
Completed | 36 (Total number of subjects completed Test drug = 74.) | 37 (Total number of subjects completed Ref drug = 73.)
Not Completed | 1 | 0
Not completed — family emergency | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: New 80 milligram (mg) atorvastatin tablets (test); marketed 80 mg atorvastatin commercial tablet (Lipitor®) (reference)
Arm/Group | Total Study Population
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC Infinity)
Description: AUCinf = Area under the plasma concentration-time curve from time 0 (predose) extrapolated to infinite time; measured in nanograms times hour per milliliter (ng*hr/mL). Pharmacokinetic (PK) parameters derived from subject's concentration data; collected Period 1, Day 1 to Day 4; Period 2, Day 1 to Day 4.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population defined as all subjects randomized and treated who had > = 1 of the parameters of primary interest in > = 1 treatment period.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Test Drug: New (test) 80 milligram (mg) atorvastatin tablets as a single dose in the first intervention period or second intervention period.
- Reference Drug: Marketed (reference) 80 mg atorvastatin commercial tablet (Lipitor®) as a single dose in the first intervention period or second intervention period.
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 74
ng*hr/mL | 168.1355 (100.77765) | 176.1731 (120.18642)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed AUCinf was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Adjusted mean difference (Test-Ref) and 90% CI was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean and 90% CI for the ratio. Alternative hypothesis of bioequivalence: (H1: θL <=µT - µR <=θU); null hypothesis of inequivalence: (Ho: µT - µR <θL or µT - µR >θU); Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was concluded if the 90% confidence intervals for the ratio of adjusted geometric means for both AUCinf and Cmax fell wholly within (80%, 125%); ANOVA; Values have been back-transformed from the log scale; Ratio of adjusted geometric means = 98.79, 90% CI [94.57 to 103.20] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means. AUClast + (Clast*/kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis

2. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Tmax = time (hours) to maximum plasma concentration (Cmax). Observed directly from data as time of first occurrence; PK parameters derived from subject's concentration data; collected Period 1, Day 1 to Day 4; Period 2, Day 1 to Day 4.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population
Measure: Median (Full Range); unit: hours
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 74
hours | 1.0 [0.5 to 4.0] | 1.0 [0.5 to 4.0]

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: AUClast = area under the plasma concentration-time curve from 0 (predose) to the time of the last measureable concentration (Clast). PK parameters derived from subject's concentration data; collected Period 1, Day 1 to Day 4; Period 2, Day 1 to Day 4.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 74
ng*hr/mL | 162.5073 (100.56590) | 170.4735 (119.70585)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed AUClast was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence interval was obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean (Test/Reference) and 90% confidence interval for the ratio; Test type: Non-Inferiority or Equivalence — Bioequivalence of the two treatments was concluded if the 90% confidence intervals for the ratio of adjusted geometric means for both AUCinf and Cmax fell wholly within (80%, 125%). AUCinf method of determination includes AUClast calculated value; ANOVA; Values have been back-transformed from the log scale; Ratio of adjusted geometric means = 98.72, 90% CI [94.41 to 103.23] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means. Log-linear trapezoidal method

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax = maximum observed plasma concentration. Measured in nanograms per milliter (ng/mL); collected Period 1, Day 1 to Day 4; Period 2, Day 1 to Day 4.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 74
ng/mL | 43.1782 (31.70609) | 43.0534 (36.47166)
Statistical Analysis 1: Comparison: Test Drug vs Reference Drug; Natural log transformed Cmax was analyzed using a mixed effects model with sequence, period and treatment as fixed effects and subject within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals were obtained from the model and exponentiated to provide estimates of the ratio of adjusted geometric mean (Test/Reference) and 90% confidence interval for the ratio; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Values have been back-transformed from the log scale; Ratio of adjusted geometric means = 104.66, 90% CI [95.73 to 114.42] — Parameter estimate = ratio (%) (test/reference) of adjusted geometric means. Observed directly from data

5. Secondary Outcome: Plasma Elimination Half-life (t1/2)
Description: t1/2 = terminal elimination half-life in hours; ln 2/kel, where kel is the termination phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression. PK parameters derived from subject's concentration data; collected Period 1, Day 1 to Day 4; Period 2, Day 1 to Day 4.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 10, 12, 24, 36, 48, 72 hours post dose
Population: PK parameter analysis population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test Drug | Reference Drug
Number analyzed (Participants) | 76 | 74
hours | 9.330 (3.1792) | 9.444 (4.0157)

ADVERSE EVENTS:
Arm/Group | Test Drug | Reference Drug
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 11/76 | 4/74
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Drug (N=76) | Reference Drug (N=74)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Dermatophytosis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 6 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.